CLINICAL TRIAL: NCT03033810
Title: FFR Versus iFR in Assessment of Hemodynamic Lesion Significance Using Gene Polymorphisms and Lesion Morphology Assessed by OCT (FiGARO Trial)
Brief Title: FFR Versus iFR in Assessment of Hemodynamic Lesion Significance
Acronym: FiGARO
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: General University Hospital, Prague (Other)
Collaborators: University of Iowa (Other)
Responsible Party: Principal Investigator, Tomas Kovarnik, The Head of Invasive Cardiology Dpt., General University Hospital, Prague
Other Study IDs: VFN_21_2016
Record Dates: First submitted 2017-01-08; First posted 2017-01-27 (Estimated); Last update posted 2017-01-27 (Estimated); Status verified 2017-01

CONDITIONS: Hemodynamics; Coronary Circulation; Tomography, Optical Coherence; Endothelial Cells; Polymorphism, Genetic

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — Genetic analysis of polymorphisms in gene for Hemoxygenase-1 and endothelial nitric oxide synthase. Patient's DNA will be isolated from peripheral blood leukocytes using standard techniques.
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (1):
- Consecutive patients with FFR and iFR: Patients with stable angina pectoris with suitable for coronary angiography will be suitable for the study
  Interventions: Device: Fractional flow reserve and instantaneous wave-free ratio

INTERVENTIONS:
Device: Fractional flow reserve and instantaneous wave-free ratio — 1. To explain discrepancies between FFR and iFR using demographic, morphological, genetic and functional indices.
  2. The development of software for the automatic detection of the lowest point of microvascular resistance.

SUMMARY:
The study will compare two invasive methods (FFR -fractional flow reserve and iFR-instantaneous wave free ratio) for assessment of hemodynamic impact of coronary stenosis on myocardial perfusion. There is a very good correlation between these methods for the assessment of hemodynamic significance in a broad spectrum of lesions. However, this correlation decreases significantly near the cut off points for each method. The investigators will try to find possible explanations for these differences by detailed morphology assessment of coronary stenosis using optical coherence tomography (OCT), analysis of gene polymorphisms that play a role in vasodilatation, and by shear stress analysis. The head-to-head comparison between FFR and iFR is not simple, because there is no "gold standard" for assessment of hemodynamic significance. Studies comparing these methods have used hyperemic stenosis resistance (HSR). For this kind of measurement it is necessary to measure the speed of blood flow. This is usually done by a Doppler analysis of flow. Unfortunately, the Doppler signal can yield many artificial or erroneous indicators, and obtaining a good quality signal is frequently time-consuming. These are the reasons that HSR has not been used in routine practice. The investigators have developed a new console and software that can provide real time analysis of the Doppler signal. It allows us to easily measure HSR, and to differentiate between the FFR and iFR measures through intrabeat analysis of microvascular resistance (lowest microvascular resistance is an essential condition for proper pressure measurement). Using this tool, it is possible to automatically identify the point of lowest microvascular resistance during each cardiac beat. The pressure gradient can then be measured at that point. This approach can eliminate almost all uncertainties in assessment of the pressure gradient produced by coronary stenosis. This tool can potentially improve the existing methods used to precisely reveal a significant stenosis. This should increase the number of hemodynamic guided procedures.

DETAILED DESCRIPTION:
BACKGROUND AND RATIONALE FOR THE STUDY Coronary artery disease (CAD) is the most frequent causes of death and disability in developed countries. The main diagnostic method for detection of CAD is a coronary angiography (CAG. However, the correlation between CAG and proven hemodynamic significance in borderline stenosis (40-70% of lumen narrowing) is only about 50%. The main method for detection of flow-limiting lesions is fractional flow reserve (FFR). FFR is calculated as distal pressure (Pd) divided by proximal pressure (Pa). The cut-off for hemodynamic significance is 0.8 and less. The use of FFR for lesion assessment has a level of recommendation of I A in European guidelines for coronary interventions from 2014. The FAME trail revealed that routine usage of FFR measurement decreased the costs of coronary interventions over two years. The reasons are smaller quantity of implanted stents and decreased number of procedures for in stent restenosis as a direct result of the lower incidence of initial stent implantation. FAME-2 trial has shown lower incidence of urgent revascularization in patients with FFR less than 0,8 treated by coronary intervention compared to those treated conservatively. This study was preliminary halted before reaching mortality endpoint for safety reasons.

Critical condition for proper FFR measurement is maximal vasodilatation. Since we do not have marker for this condition based on pressure measurement only we can only presume that it was reached by adenosine administration. There are a lot of limitations for this assumption. Foremost, technique for proper intravenous and intracoronary adenosine administration must follow strict rules and therefore can be done incorrectly and leads to wrong result in same cases. Furthermore, impaired endothelial function leads to lower response to adenosine administration. This situation can leads to false negative FFR result. The patients with CAD have frequently significant endothelial dysfunction causing lower response to vasodilatation stimuli. Endothelial dysfunction will be analyzed by a system named EndoPAT (Itamar Medical, Israel) that measures ischemia induced vasodilatation on fingers. The hypothesis that has never been tested is how polymorphism in genes for enzymes playing an important role in proper endothelial function (HO-1, hemoxygenase-1 and ENOS, endothelial NO synthase) can influences adenosine-induced vasodilatation and subsequently FFR measurement. These polymorphisms are not infrequent in population with CAD (they can be found in 40-50% in such patients).

Another possible limitation for FFR measurement is type of blood flow in coronary arteries. In presence of coronary stenosis, plaque roughness or sharp angle of a lumen the type of flow can be changed from laminar to turbulent. This type of flow is even accelerated during hyperemia induced by adenosine administration. It leads to lose of energy and exaggerates pressure drop behind stenosis that - for this reason- may not be proportional to stenosis severity. This situation can theoretically causes false positive FFR measurement. To answer this question the investigators will analyze the endothelial shear stress (ESS) that can distinguish laminar and turbulent flow and morphological indices (plaque surface, plaque eccentricity, lumen volume and lumen shape) by optical coherence tomography (OCT).

The new index able to identify physiologically significant stenosis has been recently described. It is instantaneous wave-free ratio (iFR). This technique uses a pressure gradient as well, but -unlike to FFR- iFR compares pressures (proximal and distal to stenosis) only in a specific phase of diastole (so called "wave free period"), where microvascular resistance is naturally low and stable .

The cut off point for iFR is 0.9. The correlation between FFR and iFR is between 80% and 90% in all lesions. However, the correlation between FFR and iFR close to their cut-off point is only 50%-60%. It is substantial caveat, because to estimate hemodynamic significance of borderline lesions is the main indication for these techniques. Discrepancies between FFR and iFR can be very confusing a discouraging for lesion hemodynamic assessment.

Nowadays, FFR is the only invasive method for stenosis hemodynamic assessment supported in the guidelines. However, the iFR is faster, easier and cheaper, and for these reasons it can be used for more lesions in more patients, which can improve the situation of poor penetration of hemodynamic guidance for coronary intervention in daily practice. Moreover, an increasing number of evidences implies that iFR concept can be closer to real situation in coronary arteries (avoiding non-physiologic vasodilatation). It has been shown that FFR itself has a factor of variability of 10%. This means that around the cut-off points the FFR can be just as wrong as the iFR, perhaps even more so. Moreover, the latest study has shown that iFR provides better pressure-derived diagnostic agreement with CFR (coronary flow reserve) than FFR. The investigators have been developing, in close cooperation with The University of Iowa, new technique that improves the quality of flow measurement. It was successfully tested it in a animal trial. It is a novel way of intravascular Doppler signal processing resulting in more reliable velocity curve envelope acquisition. This software improvement allows instantaneous monitoring of real time microvascular resistance during any phase of cardiac cycle. Detection of during instantaneous wave free period can serve as verification of the proprietary iFR calculation. The system may also improve iFR measurement itself, because it can measure precisely in-phase with the lowest microvascular resistance. The measurement of resistance during wave free period is named iMR (instantaneous microvascular resistance) and it has never been measured during previous trials. This index can greatly help to distinguish which method (FFR or iFR) measures the pressure gradient during lower resistance.

Further target is to develop next generation of the software that can detect lowest microvascular resistance based on pressure measurement only, without necessity of using Doppler. It could offer very precise and simple methods for hemodynamic assessment of coronary lesions. This software must be tested and verified in a human study, which will be done in the General Teaching Hospital (where both intracoronary pressure and flow will be measured). Its clinical availability will be tested and verified by the international cooperating centers (where only pressure indices, FFR and iFR will be measured). The foreign centers will also examine coronary OCT that will be sent to corelab in The University of Iowa, collect blood samples for genetic analysis that will be done in Prague and, depend on their possibilities, also endothelial dysfunction by EndoPAT.

The University of Iowa, Iowa, USA will analyze OCT measurement and perform 3D vessel reconstruction. This university has a world known team for the unique 3D reconstruction of coronary arteries based on angiography and optical coherence tomography. This institution will do an automated analysis of plaque surfaces as well.

HYPOTHESES:

1. The level of microvascular resistance can be used to distinguish which type of measurement (FFR or iFR) was done during the lower and more stable stage of microvascular resistance. This comparison can possibly explain discrepancies between FFR and iFR measurements.
2. Based on new software, using pressure measurements only, it will be possible to automatically detect the time period with the lowest microvascular resistance. This could improve accuracy of both FFR and iFR measurements.
3. Plaque ruptures, erosions, irregularities of plaque geometry and plaque located near to bifurcations cause turbulence in blood flow. This accelerated pressure drop can lead to a false positive FFR.
4. Inadequate vasodilation caused by endothelial dysfunction can lead to false negative FFR.
5. Endothelial dysfunction can be more frequently found in patients with the risk type of polymorphism in genes playing an important role in vessel vasodilatation (ENOS, HO-1)

AIMS AND EXPECTED IMPACT ON CLINICAL PRACTICE

1. To use new software (developed at the author's workplace in cooperation with The University of Iowa) to determine which of two methods for the functional assessment of coronary stenosis (FFR and iFR) perform their measurements during a lower level of microvascular resistance. This software can measure microvascular resistance in real time.
2. To develop a new version of software for the detection of microvascular resistance level, based only on intracoronary pressures without flow analysis. This could substantially improve the accuracy of both pressure-based measurements, and potentially increase the correlation between pressure based measurements and flow-based CFR.
3. To study the potential influence of endothelial dysfunction and plaque morphology on discrepancies between FFR and iFR during functional assessments of coronary stenosis.
4. To study the influence of gene polymorphisms on endothelial dysfunction

METHODS Study design Patients with stable angina pectoris with suitable for coronary angiography will be suitable for the study. We plan to include 250 patients to the study (50 from General University Hospital in Prague and 200 from cooperating centers).

Functional examinations of coronary arteries. Coronary angiography will be performed as a first procedure for detection of severity and extent of coronary atherosclerosis. Stenosis between 40-80% (based on CAG) will be suitable for morphological and functional examinations. Combo wire (Volcano Corp., USA) for pressure and flow measurement will be introduced behind the lesion and basal indices will be measured during basal flow condition: basal flow speed, pressure gradient (Pd/Pa), iFR, Pd/Pa during lowest microvascular resistance proven by Doppler analysis, iMR. Adenosine will be administered either intracoronary as a bolus (240 ug) or in continual infusion (140 μg/kg/min) based on local practice. The hyperemic indices will be measured: maximal flow speed, CFR, FFR, HSR (hyperemic stenosis resistance. Cooperating centers will perform pressure measurements (FFR, iFR, Pd/Pa) only and they will send a raw data for further analysis (off-line calculation of iFR using the new software) in General Teaching Hospital in Prague.

Morphological examinations of coronary arteries Morphological assessment of the lesions will be done by OCT (St. Jude Medical, Inc). Catheter will be placed behind stenosis. Pullback will be done during flushing of contrast dye. OCT measurement will help to choose optimal treatment strategy by proper measuring of lumen size in a lesion and in the reference segments. PCI will be done according to local practice. OCT can be use after procedure for checking results, but this second examination is not part of the study.

More detail analyze will be done from 3D vessel reconstruction in The University of Iowa that is well know center for 3D coronary reconstruction. Scientific team from this university have received two US patents for 3D coronary reconstruction.

The methodology of 3 D reconstruction of coronary arteries The two-plane angiograms will be taken immediately prior to the pullback start and cover at least one heart cycle each. They will be used to extract the catheter path automatically along the expected pullback trajectory by a dynamic programming approach. From the known imaging geometry, an accurate 3-D model of the catheter path within the respective vessel segment is generated for end-diastolic heart phase. For OCT acquisition, motorized pullback ensures a constant pullback speed, thus allowing to asses each OCT image frame a specific location on the 3-D catheter trajectory model. The relative and absolute orientations of the OCT frames will be determined using previously reported system for establishing the absolute orientation in 3-D on IVUS (intravascular ultrasound) images. Visualization will be based on automated encoding of the derived contour data in VRML (Virtual Reality Modeling Language). Quantitative data can be derived from the contour data, such as luminal dimensions and plaque-cap thickness, actually considering the vessel curvature in contrast to conventional OCT reconstruction systems. The space between adjacent contours is interpolated to form a volume element. In locations of the plaque cap, integrating over an entire vessel segment or any part thereof yields the total plaque cap volume enclosed by the inner and outer cap surfaces. The quantification values can be included into the VRML model by color per vertex encoding, thus allowing an easy and fast visual assessment of the lesion or the results of the intervention by the physician.

Endothelial shear stress analysis. A steady flow computational fluid dynamics (CFD) analysis will be performed in the reconstructed arterial segments in order to analyze for the local fluid dynamic characteristics along the vessel segment.

Examination of endothelial dysfunction. Endothelial dysfunction will be measured by a system named EndoPAT (Itamar Medical, Israel). EndoPAT uses peripheral artery tone signal (PAT) for non-invasively measuring arterial tone changes in peripheral arterial beds17.

Genetic analysis of polymorphisms in gene for HO-1 and ENOS Patient's DNA will be isolated from peripheral blood leukocytes using standard techniques.

Statistical analysis Data will be prospectively stored in a database and will be processed using the software JMP®10.0.0, Copyright © 2012 SAS (Statistical analysis software) Institute Inc. (http://www.jmp.com) in collaboration with a professional statistician.

ELIGIBILITY:
Inclusion Criteria:

* Stable angina pectoris
* Age 18-80 years
* Signed inform consent
* Coronary arteries without severe tortuosity and calcifications
* Normal blood flow in coronary arteries (TIMI flow III)
* Coronary artery stenosis less than 80% during CAG

Exclusion Criteria:

* Hemodynamic instability, cardio-pulmonary resuscitation in a same day
* Thrombosis in a target coronary artery visible during angiography
* Patients after or with planned coronary artery bypass grafting
* Severe bronchial asthma or atrio-ventricular block higher than first degree (contraindication for adenosine administration)
* Renal insufficiency with creatinine level more than 180 umol/l
* Known allergy to iodine contrast
* Pregnancy

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients with stable angina pectoris indicated for lesion hemodynamic assessment for bordeline stensois found during coronary angiography
Sampling Method: Non-Probability Sample
Enrollment: 200 (Estimated)
Dates: Start 2017-01; Primary Completion 2019-06 (Estimated); Study Completion 2019-12 (Estimated)

PRIMARY OUTCOMES:
Presence of endothelial dysfunction, plaque superficial irregularities and gene polymorphisms in patients with screpancies between FFR and iFR during functional assessments of coronary stenosis. | 2017-2019
  Endothelial dysfunction measured by EndoPAT, plaque superficial irregularities measured by OCT and gene polymorphisms in ENOS and HO-1 can be different in patients with discrepancy between FFR and iFR compared to known results from patients with coronary artery disease.

SECONDARY OUTCOMES:
To use a new software to determine which of two methods for the functional assessment of coronary stenosis (FFR and iFR) perform their measurements during a lower level of microvascular resistance. | 2017-2019
  This software will measure microvascular resistance. It´s stable and minimal value is an essential condition for precise assessment of lesion severity by pressure measurement. Lower level of microvascular resistence during FFR or iFR measurements can help to distinguish, which of these two measurements is more relyable.
To develop a new version of aforementioned software for the detection of microvascular resistance level, based only on intracoronary pressures without flow analysis | 2017-2019
  For analysis of microvascular resistance is necessary to measure coronary flow. This type of measurement is time consuming and difficult. The investigators will try to find a marker of low microvascular resistance during assessment of intracoronary pressure, which is easy to measure.

CONTACTS AND LOCATIONS:
Locations (1):
- II. interni klinika VFN, Prague, Czechia

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Park SJ, Kang SJ, Ahn JM, Shim EB, Kim YT, Yun SC, Song H, Lee JY, Kim WJ, Park DW, Lee SW, Kim YH, Lee CW, Mintz GS, Park SW. Visual-functional mismatch between coronary angiography and fractional flow reserve. JACC Cardiovasc Interv. 2012 Oct;5(10):1029-36. doi: 10.1016/j.jcin.2012.07.007. PMID 23078732
- [Background] Kern MJ, Lerman A, Bech JW, De Bruyne B, Eeckhout E, Fearon WF, Higano ST, Lim MJ, Meuwissen M, Piek JJ, Pijls NH, Siebes M, Spaan JA; American Heart Association Committee on Diagnostic and Interventional Cardiac Catheterization, Council on Clinical Cardiology. Physiological assessment of coronary artery disease in the cardiac catheterization laboratory: a scientific statement from the American Heart Association Committee on Diagnostic and Interventional Cardiac Catheterization, Council on Clinical Cardiology. Circulation. 2006 Sep 19;114(12):1321-41. doi: 10.1161/CIRCULATIONAHA.106.177276. Epub 2006 Aug 28. PMID 16940193
- [Background] Tonino PA, De Bruyne B, Pijls NH, Siebert U, Ikeno F, van' t Veer M, Klauss V, Manoharan G, Engstrom T, Oldroyd KG, Ver Lee PN, MacCarthy PA, Fearon WF; FAME Study Investigators. Fractional flow reserve versus angiography for guiding percutaneous coronary intervention. N Engl J Med. 2009 Jan 15;360(3):213-24. doi: 10.1056/NEJMoa0807611. PMID 19144937
- [Background] De Bruyne B, Fearon WF, Pijls NH, Barbato E, Tonino P, Piroth Z, Jagic N, Mobius-Winckler S, Rioufol G, Witt N, Kala P, MacCarthy P, Engstrom T, Oldroyd K, Mavromatis K, Manoharan G, Verlee P, Frobert O, Curzen N, Johnson JB, Limacher A, Nuesch E, Juni P; FAME 2 Trial Investigators. Fractional flow reserve-guided PCI for stable coronary artery disease. N Engl J Med. 2014 Sep 25;371(13):1208-17. doi: 10.1056/NEJMoa1408758. Epub 2014 Sep 1. PMID 25176289
- [Background] Kral A, Kovarnik T, Kralik L, Skalicka H, Horak J, Mintz GS, Uhrova J, Sonka M, Wahle A, Downe R, Aschermann M, Martasek P, Linhart A. Genetic variants in haem oxygenase-1 and endothelial nitric oxide synthase influence the extent and evolution of coronary artery atherosclerosis. Folia Biol (Praha). 2011;57(5):182-90. doi: 10.14712/fb2011057050182. PMID 22123460
- [Background] Meuwissen M, Chamuleau SA, Siebes M, Schotborgh CE, Koch KT, de Winter RJ, Bax M, de Jong A, Spaan JA, Piek JJ. Role of variability in microvascular resistance on fractional flow reserve and coronary blood flow velocity reserve in intermediate coronary lesions. Circulation. 2001 Jan 16;103(2):184-7. doi: 10.1161/01.cir.103.2.184. PMID 11208673
- [Background] Chatzizisis YS, Coskun AU, Jonas M, Edelman ER, Feldman CL, Stone PH. Role of endothelial shear stress in the natural history of coronary atherosclerosis and vascular remodeling: molecular, cellular, and vascular behavior. J Am Coll Cardiol. 2007 Jun 26;49(25):2379-93. doi: 10.1016/j.jacc.2007.02.059. Epub 2007 Jun 8. PMID 17599600
- [Background] Sen S, Escaned J, Malik IS, Mikhail GW, Foale RA, Mila R, Tarkin J, Petraco R, Broyd C, Jabbour R, Sethi A, Baker CS, Bellamy M, Al-Bustami M, Hackett D, Khan M, Lefroy D, Parker KH, Hughes AD, Francis DP, Di Mario C, Mayet J, Davies JE. Development and validation of a new adenosine-independent index of stenosis severity from coronary wave-intensity analysis: results of the ADVISE (ADenosine Vasodilator Independent Stenosis Evaluation) study. J Am Coll Cardiol. 2012 Apr 10;59(15):1392-402. doi: 10.1016/j.jacc.2011.11.003. Epub 2011 Dec 7. PMID 22154731
- [Background] Petraco R, van de Hoef TP, Nijjer S, Sen S, van Lavieren MA, Foale RA, Meuwissen M, Broyd C, Echavarria-Pinto M, Foin N, Malik IS, Mikhail GW, Hughes AD, Francis DP, Mayet J, Di Mario C, Escaned J, Piek JJ, Davies JE. Baseline instantaneous wave-free ratio as a pressure-only estimation of underlying coronary flow reserve: results of the JUSTIFY-CFR Study (Joined Coronary Pressure and Flow Analysis to Determine Diagnostic Characteristics of Basal and Hyperemic Indices of Functional Lesion Severity-Coronary Flow Reserve). Circ Cardiovasc Interv. 2014 Aug;7(4):492-502. doi: 10.1161/CIRCINTERVENTIONS.113.000926. Epub 2014 Jul 1. PMID 24987048
- [Background] van de Hoef TP, Nolte F, EchavarrIa-Pinto M, van Lavieren MA, Damman P, Chamuleau SA, Voskuil M, Verberne HJ, Henriques JP, van Eck-Smit BL, Koch KT, de Winter RJ, Spaan JA, Siebes M, Tijssen JG, Meuwissen M, Piek JJ. Impact of hyperaemic microvascular resistance on fractional flow reserve measurements in patients with stable coronary artery disease: insights from combined stenosis and microvascular resistance assessment. Heart. 2014 Jun;100(12):951-9. doi: 10.1136/heartjnl-2013-305124. Epub 2014 Apr 11. PMID 24727867
- [Background] Wahle A, Prause GP, von Birgelen C, Erbel R, Sonka M. Fusion of angiography and intravascular ultrasound in vivo: establishing the absolute 3-D frame orientation. IEEE Trans Biomed Eng. 1999 Oct;46(10):1176-80. doi: 10.1109/10.790492. PMID 10513120
- [Background] Wahle A, Prause PM, DeJong SC, Sonka M. Geometrically correct 3-D reconstruction of intravascular ultrasound images by fusion with biplane angiography--methods and validation. IEEE Trans Med Imaging. 1999 Aug;18(8):686-99. doi: 10.1109/42.796282. PMID 10534051
- [Background] Perktold K, Hofer M, Rappitsch G, Loew M, Kuban BD, Friedman MH. Validated computation of physiologic flow in a realistic coronary artery branch. J Biomech. 1998 Mar;31(3):217-28. doi: 10.1016/s0021-9290(97)00118-8. PMID 9645536
- [Background] Ethier CR. Computational modeling of mass transfer and links to atherosclerosis. Ann Biomed Eng. 2002 Apr;30(4):461-71. doi: 10.1114/1.1468890. PMID 12085998
- [Background] Weydahl ES, Moore JE. Dynamic curvature strongly affects wall shear rates in a coronary artery bifurcation model. J Biomech. 2001 Sep;34(9):1189-96. doi: 10.1016/s0021-9290(01)00051-3. PMID 11506789
- [Background] Bonetti PO, Pumper GM, Higano ST, Holmes DR Jr, Kuvin JT, Lerman A. Noninvasive identification of patients with early coronary atherosclerosis by assessment of digital reactive hyperemia. J Am Coll Cardiol. 2004 Dec 7;44(11):2137-41. doi: 10.1016/j.jacc.2004.08.062. PMID 15582310
- [Background] Jeremias A, Maehara A, Genereux P, Asrress KN, Berry C, De Bruyne B, Davies JE, Escaned J, Fearon WF, Gould KL, Johnson NP, Kirtane AJ, Koo BK, Marques KM, Nijjer S, Oldroyd KG, Petraco R, Piek JJ, Pijls NH, Redwood S, Siebes M, Spaan JAE, van 't Veer M, Mintz GS, Stone GW. Multicenter core laboratory comparison of the instantaneous wave-free ratio and resting Pd/Pa with fractional flow reserve: the RESOLVE study. J Am Coll Cardiol. 2014 Apr 8;63(13):1253-1261. doi: 10.1016/j.jacc.2013.09.060. Epub 2013 Nov 6. PMID 24211503
- [Background] Eshtehardi P, McDaniel MC, Suo J, Dhawan SS, Timmins LH, Binongo JN, Golub LJ, Corban MT, Finn AV, Oshinski JN, Quyyumi AA, Giddens DP, Samady H. Association of coronary wall shear stress with atherosclerotic plaque burden, composition, and distribution in patients with coronary artery disease. J Am Heart Assoc. 2012 Aug;1(4):e002543. doi: 10.1161/JAHA.112.002543. Epub 2012 Aug 24. PMID 23130168
- [Background] Campbell IC, Timmins LH, Giddens DP, Virmani R, Veneziani A, Rab ST, Samady H, McDaniel MC, Finn AV, Taylor WR, Oshinski JN. Computational Fluid Dynamics Simulations of Hemodynamics in Plaque Erosion. Cardiovasc Eng Technol. 2013 Dec;4(4):10.1007/s13239-013-0165-3. doi: 10.1007/s13239-013-0165-3. PMID 24223678
- [Background] Finet G, Huo Y, Rioufol G, Ohayon J, Guerin P, Kassab GS. Structure-function relation in the coronary artery tree: from fluid dynamics to arterial bifurcations. EuroIntervention. 2010 Dec;6 Suppl J:J10-5. doi: 10.4244/EIJV6SUPJA3. No abstract available. PMID 21930472
- [Derived] Kovarnik T, Hitoshi M, Kral A, Jerabek S, Zemanek D, Kawase Y, Omori H, Tanigaki T, Pudil J, Vodzinska A, Branny M, Stipal R, Kala P, Mrozek J, Porzer M, Grezl T, Novobilsky K, Mendiz O, Kopriva K, Mates M, Chval M, Chen Z, Martasek P, Linhart A; FiGARO trial investigators. Fractional Flow Reserve Versus Instantaneous Wave-Free Ratio in Assessment of Lesion Hemodynamic Significance and Explanation of their Discrepancies. International, Multicenter and Prospective Trial: The FiGARO Study. J Am Heart Assoc. 2022 May 3;11(9):e021490. doi: 10.1161/JAHA.121.021490. Epub 2022 May 3. PMID 35502771
- [Derived] Jerabek S, Zemanek D, Pudil J, Bayerova K, Kral A, Kopriva K, Kawase Y, Omori H, Tanigaki T, Chen Z, Vodzinska A, Branny M, Matsuo H, Mates M, Sonka M, Kovarnik T. Endothelial dysfunction assessed by digital tonometry and discrepancy between fraction flow reserve and instantaneous wave free ratio. Acta Cardiol. 2020 Aug;75(4):323-328. doi: 10.1080/00015385.2019.1586089. Epub 2019 Apr 4. PMID 30945607